CLINICAL TRIAL: NCT03405727
Title: Improvement of Sarcopenia in Sarcopenia Patients Following Two Different Diets
Brief Title: Improvement of Sarcopenia in Patients Following Two Different Diets
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of human ressources
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Tatiana Besse-Hammer, Head of clinic, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUB-diet
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment (No Intervention)
- Oral dietary supplements (Experimental)
  Interventions: Dietary Supplement: Oral dietary supplements

INTERVENTIONS:
Dietary Supplement: Oral dietary supplements — Protein enriched diet
  Arms: Oral dietary supplements

SUMMARY:
Sarcopenia is defined as a decrease in muscular strength and muscle mass, accompanied by a decrease in physical performance. Seniors might develop sarcopenia because of a decreased physical activity and a decreased protein intake. Many patients also develop sarcopenia after a long stay in an intensive care unit.

Protein intake is very important when treating sarcopenia. However, meeting the protein requirements at home proves difficult. Oral dietary supplements, given in addition to the other known recommendations, might provide a solution.

This study will assess the efficacy of the oral dietary supplements for the treatment of sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized within the CHU Brugmann, Brussels
* Patients diagnosed with sarcopenia (by means of a dynamometer)
* Patients having stayed in an intensive care unit for longer than 5 weeks

Exclusion Criteria:

* Oncology patients
* Anorexic patients
* Patients having a life expectancy of less than 6 months
* Demented patients
* BPCO patients
* Patients with neuropathies

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
Prehension force | 3 months after first consultation
  Prehension force, as measured by a dynamometer on the dominant hand
Prehension force | 6 months after first consultation
  Prehension force, as measured by a dynamometer on the dominant hand
Fat mass evaluation | 3 months after first consultation
  Measured by a Harpaden compass on the tricipital skin fold
Fat mass evaluation | 6 months after first consultation
  Measured by a Harpaden compass on the tricipital skin fold
Muscle mass evaluation | 3 months after first consultation
  Brachial muscular circumference (measured by tape)
Muscle mass evaluation | 6 months after first consultation
  Brachial muscular circumference (measured by tape)
Walking speed | 3 months after first consultation
  Walking speed on a 4 meters distance
Walking speed | 6 months after first consultation
  Walking speed on a 4 meters distance
"Time Up and Go" test | 3 months after first consultation
  Mobility assessment of the patient
"Time Up and Go" test | 6 months after first consultation
  Mobility assessment of the patient
Sedentary lifestyle questionnaire | 3 months after first consultation
  Evaluation of the physical activity by means of a questionnaire
Sedentary lifestyle questionnaire | 6 months after first consultation
  Evaluation of the physical activity by means of a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Turkan Dalgic, Principal Investigator — Haute Ecole Lucia De Brouckère
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No